CLINICAL TRIAL: NCT00448916
Title: A 12-month Open-label Extension Study Evaluating The Safety And Tolerability Of Flexible Doses Of Pregabalin In Pediatric Patients With Partial Onset Seizures
Brief Title: Open-Label Extension Study Of Safety And Tolerability Of Pregabalin In Pediatric Patients With Partial-Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081075; 2010-020731-39 (EudraCT Number)
Record Dates: First submitted 2007-03-15; First posted 2007-03-19 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2014-11

CONDITIONS: Epilepsies, Partial
Keywords: Partial-onset seizures; epilepsy; pediatric; pregabalin; 1 year extension study; safety; tolerability
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregabalin (Experimental): Orally-administered pregabalin
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — Orally-administered pregabalin

SUMMARY:
The study will evaluate the long-term safety and tolerability of pregabalin in pediatric patients, age 1 month through 16 years, with partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

* Partial onset seizures, incompletely controlled on 1-3 medications
* At least 1 seizure per 28 days, on average
* Completion of study A0081074

Exclusion Criteria:

* Primary generalized seizures
* Progressive CNS pathology
* Failure to tolerate pregabalin in study A0081074

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2007-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (16):
  - University of South Alabama, Mobile, Alabama
  - University of South Alabama Department of Neurology, Mobile, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - The Children's Clinica of Jonesboro, P.A, Jonesboro, Arkansas
  - Clinical Study Centers, L. L. C., Little Rock, Arkansas
  - UCSF Neurology Clinic, San Francisco, California
  - Child Neurology Center of Northwest Florida, Gulf Breeze, Florida
  - The Office of Sergio J Jacinto, MD, Tampa, Florida
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - St. John's Clinic, Springfield, Missouri
  - St. John's Hospital, Springfield, Missouri
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Road Runner Research, Ltd., San Antonio, Texas
- Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico
- Yonsei University College of Medicine Severance Hospital / Department of Pediatric Neurology, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081075&StudyName=Open-Label%20Extension%20Study%20Of%20Safety%20And%20Tolerability%20Of%20Pregabalin%20In%20Pediatric%20Patients%20With%20Partial-Onset%20Seizures

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was a dose extension study of pediatric participants with refractory partial-onset seizures who had completed study A0081074 (NCT00437281). Participants were enrolled in 3 countries at 13 study centers with 13 investigators: Republic of Korea (1 center), Mexico (1 center), and the United States (11 centers).
Pre-assignment Details: Each participant was restricted to the dose levels that they had previously tolerated, or that had shown acceptable safety and tolerability in study A0081074 (NCT00437281) for the participant's age group.
Groups:
- Pregabalin: 1-23 Months: Age group included 1-23 months. Pregabalin was administered orally as liquid formulation at dose of 2.5, 5, 7.5, 10, or 15 mg/kg/day for 12 Months.
- Pregabalin: 2-6 Years: Age group included 2-6 years. Pregabalin was administered orally as liquid formulation at dose of 2.5, 5, 7.5, 10, or 15 mg/kg/day for 12 Months..
- Pregabalin: 7-11 Years: Age group included 7-11 years. Pregabalin was administered orally as capsule formulation and liquid formulation was used if participants was unable to swallow capsules. Doses of 2.5, 5, 7.5, 10, or 15 mg/kg/day were given for 12 Months.
- Pregabalin: 12-16 Years: Age group included 12-16 years. Pregabalin was administered orally as capsule formulation and liquid formulation was used if participants was unable to swallow capsules. Doses of 2.5, 5, 7.5, 10, or 15 mg/kg/day were given for 12 Months.
Period: Overall Study
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Started | 16 | 15 | 12 | 11
Completed | 9 | 9 | 6 | 5
Not Completed | 7 | 6 | 6 | 6
Not completed — Adverse Event | 2 | 2 | 3 | 2
Not completed — Lack of Efficacy | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 3 | 3 | 1 | 1
Not completed — Other | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years | Total
Number analyzed (Participants) | 16 | 15 | 12 | 11 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 1.18 (0.57) | 4.14 (1.23) | 9.98 (1.30) | 14.86 (1.53) | 6.74 (5.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 5 | 3 | 25
  Male | 8 | 6 | 7 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE).
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A serious adverse event (SAE) is any untoward medical occurrence at any dose that: results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in congenital anomaly/birth defect.
Time Frame: 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  Participants with AEs | 14 | 13 | 11 | 9
  Participants with serious AEs | 8 | 3 | 0 | 1
  Participants with severe AEs | 7 | 4 | 0 | 1

2. Secondary Outcome: Number of Participants With Change From Previous Physical Examination Results at Visit 1, Week 1, Month 1, Month 6, Month 12/Early Termination and Follow-up.
Description: Changes from previous examinations in physical examination were reported. Examination of abdomen, breasts, ears, extremities, eyes, genitourinary, head, heart, lungs, lymph nodes, mouth, musculoskeletal, neck, nose, ocular fundi, skin, throat, thyroid and general examinations were done. Evaluation was done based on presence of abnormality which were noted as "abnormal" and no abnormalities in the sites were reported as "normal". Any change from the previous physical examination results were noted.
Time Frame: Visit 1, Week 1, Month 1, Month 6, Month 12/Early Termination and Follow-up.
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  Week 1 (N=16,13,11,10) | 2 | 1 | 0 | 0
  Month 1 (N=14,13,10,10) | 1 | 1 | 0 | 0
  Month 6 (N=11,10,6,7) | 1 | 1 | 0 | 0
  Month 12/Eary Termination (N=16,12,12,9) | 1 | 2 | 1 | 1
  Follow-up (N=6,4,9,6) | 0 | 0 | 1 | 0

3. Secondary Outcome: Number of Participants With Change From Previous Neurological Examination Results at Visit 1, Week 1, Month 1, Month 6, Month 12/Early Termination and Follow-up.
Description: Changes from previous examinations in neurological examination were reported. The neurologic exam were performed by a pediatric neurologist or qualified staff member. Coordination, cranial nerves, gait, level of consciousness, lower and upper extremity sensation, muscle strength, muscle tone, nystagmus, reflexes, Romberg test, and speech were examined.
Time Frame: Visit 1, Week 1, Month 1, Month 6, Month 12/Early Termination and Follow-up
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Groups:
- Pregabalin: 12-16 Years: Age group included 12-16 years. Pregabalin was administered orally as liquid or capsule formulation at dose of 2.5, 5, 7.5, 10, or 15 mg/kg/day.
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  Week 1 (N=16,13,11,10) | 1 | 0 | 0 | 0
  Month 1 (N=14,13,10,10) | 0 | 0 | 0 | 0
  Month 6 (N=11,10,6,7) | 0 | 0 | 0 | 0
  Month 12/Early Termination (N=16,11,12,9) | 0 | 0 | 0 | 0
  Follow-up (N=6,4,9,6) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Significant Change in Supine Diastolic Blood Pressure (BP) at Post-Baseline Visits (Visit 1 to 12 Months).
Description: Participants with significant supine diastolic BP values with the criteria ≥ 20% increase from Baseline or ≥ 20% decrease from Baseline or > 1.25 times upper limit of normal (ULN) or < 0.9 times lower limit of normal (LLN) were identified and recorded. The categorical summary of Post-Baseline supine diastolic BP data are presented below.
Time Frame: Visit 1 to 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  ≥ 20% increase from Baseline | 12 | 5 | 8 | 3
  ≥ 20% decrease from Baseline | 5 | 7 | 3 | 3
  > 1.25 * ULN | 1 | 1 | 0 | 0
  < 0.9 * LLN | 0 | 0 | 3 | 0

5. Secondary Outcome: Number of Participants With Significant Change in Supine Systolic BP at Post Baseline Visits (Visit 1 to 12 Months).
Description: Participants with significant supine systolic BP values with the criteria ≥ 30% increase from Baseline or ≥ 30% decrease from Baseline or > 1.25 times ULN or < 0.9 times LLN were identified and recorded. The categorical summary of Post-Baseline supine systolic BP data are presented below.
Time Frame: Visit 1 to 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  ≥ 30% increase from Baseline | 2 | 3 | 1 | 1
  ≥ 30% decrease from Baseline | 2 | 1 | 0 | 0
  > 1.25 * ULN | 0 | 0 | 0 | 0
  < 0.9 * LLN | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Significant Change in Supine Heart Rate (HR) at Post Baseline Visits (Visit 1 to 12 Months).
Description: Participants with significant heart rate values with the criteria > 1.5 times ULN or < 0.9 times LLN were identified and recorded. The categorical summary of Post-Baseline supine HR data are presented below.
Time Frame: Visit 1 to 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  > 1.5 * ULN | 0 | 0 | 0 | 0
  < 0.9 * LLN | 5 | 2 | 1 | 0

7. Secondary Outcome: Derived Body Mass Index Data (BMI) at Month 12/Early Termination.
Description: BMI was calculated from height and weight measured at Month 12 visit using the formula: weight(kg)/height(m)2.
Time Frame: Month 12/Early Termination
Population: Safety analysis set: All participants who received at least one dose of study medication were included. Data was available for 15, 11, 10 and 7 participants in Pregabalin 1-23 months group, 2-6 years group, 7-11 years group and 12-16 years group respectively.
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 15 | 11 | 10 | 7
Kg/m^2 | 16.2 (1.73) | 18.0 (3.52) | 20.6 (6.52) | 24.8 (7.72)

8. Secondary Outcome: Change From Baseline in Body Weight at Day 9, Week 1, Month 1, Month 2, Month 4, Month 6, Month 9, Month 12/Early Termination and Follow-up.
Description: Weight was recorded in kilograms and weight change from Baseline was reported.
Time Frame: Baseline, Day 9, Week 1, Month 1, Month 2, Month 4, Month 6, Month 9, Month 12/Early Termination and Follow-up
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Kg
  Day 9 (N=16,14,12,11) | 0.1 (0.16) | 0.1 (0.29) | -0.1 (0.79) | 0.4 (1.07)
  Week 1 (N=16,13,11,10) | 0.3 (0.29) | 0.4 (0.61) | 1.5 (1.15) | 1.2 (1.43)
  Month 1 (N=14,13,10,10) | 0.4 (0.45) | 0.8 (0.73) | 2.1 (1.77) | 2.4 (1.52)
  Month 2 (N=11,12,8,9) | 1.0 (0.73) | 1.2 (1.12) | 3.8 (3.25) | 3.0 (1.81)
  Month 4 (N=11,10,7,9) | 1.3 (0.86) | 1.3 (1.29) | 5.2 (4.32) | 4.1 (2.28)
  Month 6 (N=11,10,6,7) | 1.8 (0.98) | 1.4 (1.52) | 5.9 (4.17) | 5.9 (3.32)
  Month 9 (N=9,10,6,5) | 2.4 (1.18) | 2.3 (2.52) | 6.3 (4.66) | 7.3 (4.32)
  Month 12/Early Termination (N=15,12,11,8) | 1.8 (1.33) | 2.4 (2.71) | 6.0 (4.78) | 6.6 (4.51)

9. Secondary Outcome: Height at Month 12/Early Termination.
Description: Height was recorded in centimeters.
Time Frame: Month 12/Early Termination
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 15 | 11 | 10 | 7
cm | 83.3 (8.87) | 109.9 (12.76) | 145.6 (13.21) | 167.3 (8.18)

10. Secondary Outcome: Number of Participants With Changes in Electrocardiogram (ECG) Data Post-Baseline Visits (Week 1 to 12 Months).
Description: Based on the criteria for safety values of potential clinical concern, the PR interval (≥200 msec; ≥25% increase from Baseline; ≥50% increase from Baseline), QRS complex (≥200 msec; ≥25% increase from Baseline), QT (≥500 msec), maximum QTcB interval (450-<480; 480-<500; ≥500 msec) and maximum QTcF interval (450-<480; 480-<500; ≥500 msec) values were calculated.
  Baseline was defined as Day 1 of the parent study A0081074 (NCT00437281). Categorical data of the Post-Baseline vists are represented below.
Time Frame: Week 1 to 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  PR interval: ≥ 200 msec | 0 | 0 | 0 | 0
  PR interval: ≥50% increase from Baseline | 0 | 0 | 0 | 0
  PR interval: ≥25% increase from Baseline | 1 | 0 | 1 | 0
  QRS interval: ≥ 200 msec | 0 | 0 | 0 | 0
  QRS interval: ≥25% increase from Baseline | 0 | 0 | 0 | 0
  QT interval: ≥ 500 msec | 0 | 0 | 0 | 0
  QTcB interval: 450-<480 msec | 1 | 1 | 1 | 2
  QTcB interval: 480-<500 msec | 0 | 0 | 0 | 0
  QTcB interval: ≥ 500 msec | 0 | 0 | 0 | 0
  QTcF interval: 450-<480 msec | 0 | 0 | 0 | 0
  QTcF interval: 480-<500 msec | 0 | 0 | 0 | 0
  QTcF interval: ≥ 500 msec | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Hematotolgical Abnormalities.
Description: Based on criteria for safety values of potential clinical concern, the participants with abnormal values were noted. Some of the values are: platelets (10*3/mm*3): <0.5 LLN or >1.75 ULN; white blood cell (WBC) count (X10E9/L): <0.6 LLN or >1.5 ULN; lymphocytes-Abs (10*3/mm*3): <0.8 LLN or >1.2 ULN; total neutrophils-Abs (10*3/mm*3): <0.8 LLN or >1.2 ULN; and eosinophils-Abs: >1.2 ULN.
Time Frame: 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  Platelets: <0.5xLLN (N=16,15,12,11) | 1 | 1 | 0 | 0
  Platelets: >1.75xULN (N=16,15,12,11) | 1 | 0 | 0 | 0
  WBC count: <0.6xLLN (N=15,15,12,11) | 1 | 2 | 0 | 0
  WBC count: >1.5xULN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Lymphocytes-Abs: <0.8xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Lymphocytes-Abs: >1.2xULN (N=15,15,12,11) | 1 | 0 | 0 | 2
  Total neutrophils-Abs: <0.8xLLN (N=15,15,12,11) | 3 | 4 | 3 | 3
  Total neutrophils-Abs: >1.2xULN (N=15,15,12,11) | 1 | 1 | 0 | 0
  Eosinophils-Abs: >1.2xULN (N=15,15,12,11) | 3 | 1 | 1 | 0
  Hemoglobin: <0.8xLLN(N=15,15,12,11) | 0 | 0 | 0 | 0
  Hematocrit: <0.8xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Red blood cell count: <0.8xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Basophils: >1.2xULN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Monocytes: >1.2xULN (N=15,15,12,11) | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Abnormalities in Urinalysis (Dipstick/Microscopy).
Description: Based on criteria for safety values of potential clinical concern, the participants with abnormal values were noted. Participants with Urine Protein (mg/dL) abnormalities (≥1) were noted based on urinalysis (dipstick). No participants with abnormalities in urinalysis (microscopy) were noted.
Time Frame: 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 11 | 15 | 11 | 11
Participants | 1 | 1 | 0 | 1

13. Secondary Outcome: Number of Participants With Abnormalities in Endocrine Panel (Hormones).
Description: Based on criteria for safety values of potential clinical concern, the participants with abnormal values were noted. Some of the criteria are: Free thyroxine (T4 free) (ng/dL): <0.8 LLN or >1.2 ULN and Thyroid-stimulating hormone (TSH) (mu/L): <0.8 LLN or >1.2 ULN.
Time Frame: 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants
  T4 (free): <0.8xLLN (N=13,13,11,10) | 0 | 1 | 0 | 0
  T4 (free): >1.2xULN (N=13,13,11,10) | 0 | 0 | 0 | 0
  TSH: <0.8xLLN (N=14,12,11,10) | 1 | 0 | 0 | 0
  TSH: >1.2xULN (N=14,12,11,10) | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Abnormalities in Creatine Kinase.
Description: Based on criteria for safety values of potential clinical concern, the participants with abnormal values in creatine kinase (>2.0 times upper limit of the reference range) (u/L) were noted.
Time Frame: 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 15 | 15 | 12 | 11
Participants | 0 | 1 | 1 | 4

15. Secondary Outcome: Seizure Frequency.
Description: Twenty-eight-day seizure frequencies were to be calculated from the seizure diaries and were to be reviewed. However, due to the nature of the data collection and due to unability to clearly differentiate no seizures versus seizures, accurate computation of this data was not performed. Hence, the seizure data was reported as AE.
Time Frame: 28 Days
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 16 | 15 | 12 | 11
Participants | NA — Due to the nature of the data collection and due to unability to clearly differentiate no seizures versus seizures, accurate computation of this data was not performed | NA — Due to the nature of the data collection and due to unability to clearly differentiate no seizures versus seizures, accurate computation of this data was not performed | NA — Due to the nature of the data collection and due to unability to clearly differentiate no seizures versus seizures, accurate computation of this data was not performed | NA — Due to the nature of the data collection and due to unability to clearly differentiate no seizures versus seizures, accurate computation of this data was not performed

16. Secondary Outcome: Number of Participants With Abnormalities in Chemistry (Including Liver Function, Renal Function, Lipids, Electrolytes, Glucose, Insulin Like Growth Factor (IGF) and IGF Binding Protein).
Description: Based on criteria for safety values of potential clinical concern, the participants with abnormal values in liver function tests, renal function tests, lipid profile, electrolytes, glucose, Insulin like growth factor (IGF) and IGF binding protein were noted and reported in this section.
Time Frame: 12 Months
Population: Safety analysis set: All participants who received at least one dose of study medication were included.
Measure: Number; unit: Participants
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years
Number analyzed (Participants) | 15 | 15 | 12 | 11
Participants
  Alanine Aminotransferase: >3.0xULN (N=15,15,12,11) | 0 | 1 | 1 | 0
  Blood Urea Nitrogen: >1.3xULN | 2 | 5 | 1 | 0
  Albumin: <0.8xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Albumin: >1.2xULN (N=15,15,12,11) | 2 | 0 | 0 | 0
  Potassium: <0.9xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Potassium: >1.1xULN (N=15,15,12,11) | 1 | 0 | 1 | 0
  Magnesium: <0.9xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Magnesium: >1.1xULN (N=15,15,12,11) | 1 | 2 | 0 | 1
  Phosphate: <0.8xLLN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Phosphate: >1.2xULN (N=15,15,12,11) | 0 | 1 | 1 | 0
  Bicarbonate (venous): <0.9xLLN (N=15,15,12,11) | 9 | 11 | 7 | 3
  Bicarbonate (venous): >1.1xULN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Glucose: <0.6xLLN (N=15,15,12,11) | 1 | 1 | 0 | 0
  Glucose: >1.5xULN (N=15,15,12,11) | 0 | 0 | 0 | 0
  Insulin-like GrowthFactor:<0.9xLLN(N=12,13,11,10) | 0 | 0 | 1 | 0
  Insulin-like GrowthFactor:>1.1xULN(N=12,13,11,10) | 5 | 8 | 4 | 6
  IGF Binding Protein: <0.9xLLN (N=12,13,11,10) | 0 | 0 | 0 | 0
  IGF Binding Protein: >1.1xULN (N=12,13,11,10) | 4 | 2 | 5 | 0
  Lipid profile cholesterol/triglycerides(N=1,4,0,1) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Visit 1 to Visit 9 (Follow-up visit)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Groups:
- Overall: This arm summarizes the AE data from all the treatment groups.
Arm/Group | Pregabalin: 1-23 Months | Pregabalin: 2-6 Years | Pregabalin: 7-11 Years | Pregabalin: 12-16 Years | Overall
Serious Adverse Events (participants affected / at risk) | 8/16 | 3/15 | 0/12 | 1/11 | 12/54
Other Adverse Events (participants affected / at risk) | 14/16 | 13/15 | 11/12 | 9/11 | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin: 1-23 Months (N=16) | Pregabalin: 2-6 Years (N=15) | Pregabalin: 7-11 Years (N=12) | Pregabalin: 12-16 Years (N=11) | Overall (N=54)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 3 | 0 | 0 | 0 | 3
Status epilepticus (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Unresponsive to stimuli (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin: 1-23 Months (N=16) | Pregabalin: 2-6 Years (N=15) | Pregabalin: 7-11 Years (N=12) | Pregabalin: 12-16 Years (N=11) | Overall (N=54)
Cyclic neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 2
Astigmatism (Eye disorders) | 1 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1 | 0 | 0 | 2
Excessive eye blinking (Eye disorders) | 0 | 0 | 1 | 0 | 1
Hypermetropia (Eye disorders) | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 3
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 1 | 1 | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 0 | 0 | 6
Faeces pale (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 3
Retching (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 4
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Crying (General disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
Irritability (General disorders) | 3 | 0 | 0 | 0 | 3
Pyrexia (General disorders) | 9 | 3 | 0 | 3 | 15
Thirst (General disorders) | 0 | 0 | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 4 | 1 | 0 | 5
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 0 | 3
Otitis media (Infections and infestations) | 4 | 4 | 0 | 0 | 8
Otitis media acute (Infections and infestations) | 2 | 1 | 0 | 0 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 2 | 1 | 0 | 3
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 1 | 0 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 2 | 0 | 10
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Anal injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Anticonvulsant drug level increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 1 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1 | 3 | 1 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 2 | 0 | 1 | 3
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 1 | 4
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Anger (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Dissociation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Dysphemia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Dyssomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 2
Personality change (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 3
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 3
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Adenoidectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.